CLINICAL TRIAL: NCT02549521
Title: Magnesium Supplementation in Elderly Females
Brief Title: Mg Induced Changes From Day 0 to Day 28 on Serum and Urine Bone Metabolic Parameters in 70 y Old Females (no 50).
Acronym: parathormon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Nycomed (Industry)
Responsible Party: Principal Investigator, Thomas Bøhmer, Prof. em., Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Nycomed 06.09.05; Nycomed contract 06.09.05 (Other Grant/Funding Number: Nycomed); Etical commitee, 548-05-99010 (Other: REK); Data inspectorate 13433 (Registry Identifier: Datatilsynet)
Record Dates: First submitted 2014-11-22; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Unspecified Disorder of Bone Density and Structure
Keywords: calcium; magnesium; vitamin D; bone turnover markers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral magnesium substitution (Active Comparator): Daily 240 mg Magnesium Nycomed Pharma. Intervention day 0 - day 28.
  Interventions: Dietary Supplement: Oral magnesium substitution
- Magnesium + or Magnesium - (Placebo Comparator): Placebo tablets without magnesium.
  Interventions: Dietary Supplement: Placebo tablets without magnesium

INTERVENTIONS:
Dietary Supplement: Oral magnesium substitution — The elderly was given tablets two times daily with calsium and vitamin D. They were further given magnesium tablets 120 mg two times daily for 28 days.
  Arms: Oral magnesium substitution
Dietary Supplement: Placebo tablets without magnesium — The elderly was given tablets two times daily with calsium and vitamin D. They were further given placebo without magnesium two times daily for 28 days.
  Arms: Magnesium + or Magnesium -

SUMMARY:
Calcium and vitamin D substitution has for a long time been used to improve osteoporosis.The main storage place for magnesium is in the bone. Magnesium is direct under calcium in the periodic system making it possible to interact with the crystal structure. Some small studies have shown beneficial effects of magnesium substitution on osteoporosis. Evidence has shown improvement with calcium, alcohol, fruit and vegetable nutrients on bone loss. It has been uncertain however, which of these factors can contribute to such a change. The effect of magnesium substitution 240 mg daily as therefore studied in two parallel groups where both received calcium carbonate 1000 mg/day and cholecalciferol 10 ug/day, one got placebo and the other received magnesium. This was studied on various expressions for bone metabolism after zero, seven and 28 days in elderly females aged 70 years old.

DETAILED DESCRIPTION:
Elderly 70 year old ladies who had been to an outpatient X-ray investigation were invited to participate in this study. They were all healthy without any signs of osteoporosis, or fractures.They were stimulated to participate by having done bone density measurements free. Patients who had used biphosphonates, oestrogens, glucocorticoids , diuretics, immunomodulating agents, or prolonged use of heparin were excluded.

Patients with possible secondary osteoporosis due to primary hyperthyroidism or chronic lung disease were also excluded. The participants were randomized into placebo or Mg-treatment groups. They were seen by the dietician, and blood and urine samples were taken at day 0, 7 and 28 at the same time these days. Medicine was prepacked for intake twice daily. They received medicine for 30 days and should only take for 28 days. The number of tablets which should be left was controlled the last day. The participants were informed about the results of the bone density measurements taken the first and the last day. All the patient contacts were undertaken by the same dietician.

ELIGIBILITY:
Inclusion Criteria:

Homeliving healthy female volunteers aged 70 years old were recruited by phone.

Exclusion Criteria:

Persons who had used:

* biphosphonates,
* oestrogens,
* glucocortocoids,
* antiepileptic drugs,
* diuretics,
* immunmodulating agents,
* prolonged usage of heparin.
* patients with possible secondary osteoporosis and
* diagnosis as:

  * inflammatory bowel disease,
  * primary hyperthyroidisms,
  * chronic obstructive lung disease

Ages: 70 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Mg induced changes from day 0-28 on serum Ca and serum Mg, (mmol/L) | 28 days
Mg induced changes from day 0-28 on ratio U Ca/creatinin and ratio of Mg/creatinin, (umol/umol) | 28 days
Mg induced changes from day 0-28 on s-calcidiol (nmol/L) | 28 days
Mg induced changes from day 0-28 on s-calcitriol (pmol/L) | 28 days
Mg induced changes from day 0-28 on s-PTH ( pmol/L) | 28 days
Mg induced changes from day 0-28 on s-Bone ALP (u/L) | 28 days
Mg induced changes from day 0-28 on s-osteocalcin (nmol/L) | 28 days
Mg induced changes from day 0-28 on s- 1-CTP (ug/L) | 28 days
Mg induced changes from day 0-28 on U-PYD/creatinin (nmol/mmol) | 28 days
Mg induced changes from day 0-28 on U-1NTx (nmol/BCE/mmol/L creatinin) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bøhmer, MD, PhD., Principal Investigator — University Hospital, Aker